CLINICAL TRIAL: NCT05039203
Title: The Risk of Symptomatic Bacteriuria and Persistence of Asymptomatic Bacteriuria After Removal of an Indwelling Urinary Catheter- a Prospective Observational Study Among Elderly Inpatients.
Brief Title: Bacteriuria and Indwelling Urinary Catheter.
Status: Active, not recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ann Tammelin, MD, Associate Professor, Region Stockholm
Other Study IDs: 2021-02410
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Bacteriuria Asymptomatic; Urinary Tract Infections
Keywords: Urinary Catheter
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples for culture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Inpatients with an indwelling urinary catheter (IUC) at admission to a rehabilitation clinic for persons ≥65 years in Sweden. Intervention is removal of the IUC.
  Interventions: Device: Indwelling urinary catheter
- Control group: Inpatients without an IUC at admission to a rehabilitation clinic for persons ≥65 years in Sweden

INTERVENTIONS:
Device: Indwelling urinary catheter — Removal of indwelling urinary catheter
  Groups: Intervention group

SUMMARY:
Investigation of 1. The incidence of symptomatic bacteriuria during four weeks after removal of an IUC in inpatients at a rehabilitation clinic for patients ≥ 65 years compared with the incidence of symptomatic bacteriuria among inpatients not treated with an IUC and 2. For how long does ABU persist in inpatients at a rehabilitation clinic for patients

≥ 65 years during a follow-up time of four weeks after IUC-removal?

ELIGIBILITY:
Inclusion Criteria:

* Admission to a rehabilitation clinic for patients ≥ 65 years in Stockholm County, Sweden
* Ability to understand oral and written instructions in Swedish
* Ability to produce a voided urine-sample

Exclusion Criteria:

* Severe cognitive failure and/or disability to understand oral and written instructions in Swedish according to the healthcare-personnel's judgment at the ward
* End-of-life care
* Physical disability to produce voided urine-samples
* Ongoing antimicrobial treatment for symptomatic bacteriuria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to a rehabilitation clinic for patients ≥ 65 years in Stockholm County, Sweden.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Symptomatic bacteriuria (urinary tract infection) | Four weeks
  Clinical diagnosis of urinary tract infection by a physician

SECONDARY OUTCOMES:
Asymptomatic bacteriuria (ABU) | One day
  Prevalence of ABU at the point of removal of an IUC compared with patients without IUC
Persistence of ABU | Four weeks
  For how long does ABU persist after IUC-removal

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Geriatric Department, Södertälje Hospital, Södertälje
  - Geriatric Department, Danderyd Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kulbay A, Joelsson-Alm E, Amilon K, Tammelin A. Asymptomatic bacteriuria and urinary tract infection in geriatric inpatients after indwelling urinary catheter removal: a descriptive two-centre study. Infect Prev Pract. 2024 Oct 24;6(4):100411. doi: 10.1016/j.infpip.2024.100411. eCollection 2024 Dec. PMID 39583881